CLINICAL TRIAL: NCT04408456
Title: Efficacy of Hydroxychloroquine (HCQ) as Post Exposure Prophylaxis (PEP) for Prevention of COVID-19 in Asymptomatic Individual at Risk for SARS-CoV-2 Infection-A Open Level Control Clinical Trial
Brief Title: Efficacy of Hydroxychloroquine (HCQ) as Post Exposure Prophylaxis (PEP) for Prevention of COVID-19
Acronym: PEP-CQ
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Deba Prasad Dhibar, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IEC-04/2020-1624
Record Dates: First submitted 2020-05-24; First posted 2020-05-29 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: CoVID-19
Keywords: CoVID-19; SARS-CoV-2; Hydroxychloroquine (HCQ); post exposure prophylaxis (PEP)
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post Exposure Prophylaxis (PEP) Group (Active Comparator): Standard therapy in the form of home quarantine for 2 weeks along with social distancing and personal hygiene Plus Tablet HCQ 400 mg q 12 hourly on day one followed by 400 mg once weekly for 3 weeks (total cumulative dose of 2000 mg)
  Interventions: Drug: HCQ; Other: Standard therapy
- Control Group (Other): Standard therapy in the form of home quarantine for 2 weeks along with social distancing and personal hygiene
  Interventions: Other: Standard therapy

INTERVENTIONS:
Drug: HCQ — Tablet HCQ 400 mg q 12 hourly on day one followed by 400 mg once weekly for 3 weeks (total cumulative dose of 2000 mg)
  Arms: Post Exposure Prophylaxis (PEP) Group
Other: Standard therapy — Home quarantine for 2 weeks plus social distancing plus personal hygiene

SUMMARY:
Novel corona virus (SARS-CoV-2) epidemic which stared from Wuhan in China is now a well established pandemic worldwide. After Italy, Spain, Germany, United Kingdom and USA, India is at the edge of becoming the next epicentre of this Pandemic. If adequate preventive and therapeutic measures are not taken, India has very high risk of affecting million of people with high mortality because of the large population along with very high population density. At present there are no definitive therapeutic drugs or vaccine are available for the treatment and prevention of SARS-CoV-2 infection. Symptomatic and supportive care are being given to COVID-19 cases along with isolation and quarantine measure are being taken for the suspected individual at risk for COVID-19 to limit the spread of the SARS-CoV-2 infection . Among the all the drugs being used for the treatment of COVID-19, hydroxychloroquine (HCQ), has given some rays of hope to battle against this deadly pandemic. HCQ has some anti viral effect against SARS-CoV in vitro. HCQ is quite safe and being used in rheumatology patients for lifelong without much side effect, so it allow for higher dose without any significant side effects and drug-drug interaction. Recently published clinical trial suggested HCQ can be used for the therapeutic purpose of the SARS-CoV-2 infection. Indian council of medical research (ICMR) has advised for HCQ prophylaxis for all asymptomatic health care workers involved in taking care of suspected or confirmed COVID-19 cases and all asymptomatic household contacts of labarotory confirmed COVID-19 cases. But there is still lack of significant scientific data to prove or disprove the efficacy of HCQ for the treatment and post exposure chemo-prophylaxis for SARS-CoV-2 infection. Being a tertiary care centre we are catering many states which include Punjab, hariyana, himachal Pradesh, Uttara khand, Uttar Pradesh. Among this Punjab have highest population of non residential Indian (NRI) and most of them have returned home. This put our institute to handle highest burden of suspected cases of SARS-CoV-2 in northern India. So we have planned this open level control clinical trial to evaluate the efficacy of post exposure prophylaxis (PEP) with HCQ for the prevention of COVID-19 in asymptomatic individuals who are at risk for SARS-CoV-2 infection. All asymptomatic individuals who have undertaken international travel in last 2 weeks and all asymptomatic individual with direct contact with laboratory confirmed cases will be advised for home quarantine for 2 weeks along with social distancing and personal hygiene. They will be given the option for taking HCQ prophylaxis. These quarantined asymptomatic individuals will be assigned into one post exposure prophylaxis (PEP) group and one control group as per inclusion and exclusion criteria. Individual who will not give consent for HCQ prophylaxis and those with contraindication for HCQ therapy like, hypersensitivity to HCQ or 4-aminoquinolone derivatives, patients with known retionopathy, cardiac arrhythmia, G6PD deficiency, psoriasis and pregnancy will be directly included in the control group. All symptomatic individual, and all health care workers related to suspected or proven COVID-19 will be excluded from the study. The PEP group will receive tablet HCQ 400 mg q 12 hourly on day one followed by 400 mg once weekly for 3 weeks (total cumulative dose of 2000 mg). The control group will not receive HCQ. Both the groups will receive standard care of therapy in the form of home quarantine for 2 weeks along with social distancing and personal hygiene. They will be followed up for 4 weeks telephonically or physically as and when required and will be enquired regarding development of any COVID-19 symptoms like fever, cough, sore throat, shortness of breath, diarrhoea, myalgia.During follow up nasopharyngeal and or throat swab of the participants will be taken for processing reverse transcription polymerase chain reaction (RTPCR) for the detection SARS-Cov-2 RNA to confirm CoVID-19. Samples for RTPCR will be taken when any asymptomatic participants become symptomatic and by the 5-14 days of contact in asymptomatic participants through in-hospital visit at the institute's communicable disease ward isolation. The participant with RTPCR positive and with or without symptoms will be defined as definite COVID-19 case and the RTPCR negative symptomatic participant will be defined as probable COVID-19 case. Asymptomatic participants with negative RTPCR will be defined as non-COVID case. Incidence of COVID-19 or probable COVID-19 or non-COVID case in previously asymptomatic participants will be compared between the PEP and control groups.

DETAILED DESCRIPTION:
Background and rational of the study:

Novel corona virus (SARS-CoV-2) epidemic which stared from Wuhan in China is now a well established pandemic worldwide affecting more than 3 lakh people with more than 15000 mortality. As Italy, Spain, Germany, United Kingdom and USA have taken over from China in term of highest burden of mortality, India is at the edge of becoming the next epicentre of this Pandemic. Presently there are around 500 active cases of corona virus disease-19 (COVID-19) in India with unfortunate mortality of 8 patients as on 24th March 2020. The clinical presentation of the COVID-19 varies from asymptomatic cases and mild symptoms of fever, cough, sore throat, headache, myalgia, nasal congestion, diarrhea to severe pneumonia, acute respiratory distress syndrome (ARDS) requiring mechanical ventilation and even multi-organ dysfunction syndrome (MODS), sepsis leading to death. If adequate preventive and therapeutic measures are not taken, India has very high risk of affecting million of people with high mortality because of the large population along with very high population density. At present there are no definitive therapeutic drugs or vaccine are available for the treatment and prevention of SARS-CoV-2 infection. Symptomatic and supportive care are being given to COVID-19 cases along with isolation and quarantine measure are being taken for the suspected individual at risk for COVID-19 to limit the spread of the SARS-CoV-2 infection.

Presently many scientist and doctors are recommending many existing available drugs (Ribavirin, lopinavir, Remdesivir, chloroquine, hydroxychloroquine) for SARS-CoV-2 infection for therapeutic and as well as prophylactic purpose . Among which hydroxychloroquine sulphate (HCQ), a chloroquine analogue has given some rays of hope to battle against this deadly pandemic. In a in vitro study researchers have found that HCQ has some anti viral effect against SARS-CoV through mechanism targeted at the host cell. HCQ is quite safe drugs as it is being used in rheumatology patients for lifelong therapy without much side effect, so it allow for higher dose without any significant side effects and drug-drug interaction. Recently published clinical trial suggested HCQ can be used for the therapeutic purpose of the SARS-CoV-2 infection and many governments including USA and India have already endorse that due to lack of any other better alternative drugs. ICMR has advised for HCQ prophylaxis for the people who are at risk for developing SARS-CoV-2 infection, all asymptomatic health care workers involved in taking care of suspected or confirmed COVID-19 cases and all asymptomatic household contacts of labarotory confirmed COVID-19 cases. But there is still lack of significant scientific data to prove or disprove the efficacy of HCQ for the treatment and post exposure chemo-prophylaxis for SARS-CoV-2 infection management. Being a tertiary care centre we are catering many states which include Punjab, hariyana, himachal Pradesh, Uttara khand, Uttar Pradesh. Among this Punjab have highest population of non residential Indian (NRI) and most of them have returned home. This put our institute to handle highest burden of suspected cases of SARS-CoV-2 in northern India. So we have planned this randomised control clinical trial to evaluate the efficacy of post exposure prophylaxis (PEP) with HCQ for the prevention of COVID-19 in asymptomatic population who are at risk for SARS-CoV-2 infection. As a research institute of national as well as international interest, it is a great opportunity for us to produce such a robust data which can be utilized in reforming national and international guidelines for the battle against of COVID-19 pandemic.

Details of method:

Aims of the study: To evaluate the efficacy of post exposure prophylaxis (PEP) with HCQ for the prevention of COVID-19 in asymptomatic individual who are at risk for SARS-CoV-2 infection.

Site of Study: The study will be conducted in the special screening OPD for the SARS-CoV-2 at Emergency and medical outpatient department (EMOPD & MOPD) and Communicable disease ward of the Post Graduate Institute of Medical Education and Research (PGIMER), Chandigarh, India. The study will be done under the collaboration of the department of Internal Medicine, Virology and Pharmacology of the institute, PGIMER,Chandigarh.

Study Design: It is an open label controlled clinical trial. The study will be done in two groups. After screening of the suspected SARS-CoV-2 infected individuals, asymptomatic quarantined individuals will be assigned into two study groups. Post exposure prophylaxis (PPE) group will receive tablet HCQ 400 mg q 12 hourly on day one followed by 400 mg once weekly for 3 weeks (total cumulative dose of 2000 mg). The control group will not receive HCQ. Both the groups will receive standard care of therapy. Individual who will not give consent for HCQ prophylaxis and those with contraindication for HCQ therapy will be directly included in the control group. They will be followed up for 4 weeks telephonically or physically as and when required.

Screening and Enrolment of Patients: All the suspected cases of COVID-19 will be screened as per ICMR guideline at special screening OPD for the SARS-CoV-2 at Emergency and medical outpatient department (EMOPD & MOPD. All asymptomatic individuals who have undertaken international travel in last 2 weeks and all asymptomatic individual with direct contact with laboratory confirmed cases will be advised for home quarantine for 2 weeks along with social distancing and personal hygiene. They will be given the option for taking HCQ prophylaxis. They will be assigned into one post exposure prophylaxis (PEP) group and one control croup as per inclusion and exclusion criteria after getting informed consent.Individual who will not give consent for HCQ prophylaxis and patients with contraindication for HCQ therapy like, hypersensitivity to HCQ or 4-aminoquinolone derivatives, patients with known retionopathy, cardiac arrhythmia, G6PD deficiency, psoriasis and pregnancy will be directly included in the control groups.

ELIGIBILITY:
Inclusion:

1. Asymptomatic individuals who have undertaken International travel in last 2 weeks
2. Asymptomatic individual with direct contact with laboratory confirmed cases

Exclusion:

1. Symptomatic individual
2. Health care worker

Individual who will not give consent for HCQ prophylaxis and patients with contraindication for HCQ therapy like, hypersensitivity to HCQ or 4-aminoquinolone derivatives, patients with known retionopathy, cardiac arrhythmia, G6PD deficiency, psoriasis and pregnancy will be directly included in the control groups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence confirmed case of COVID-19 | 3 weeks
  Participant with RTPCR positive for SARS-CoV-2 and with or without symptoms will be defined as definite COVID-19 case.
Incidence of probable case of COVID-19 | 3 weeks
  The participant with new onset symptoms, but RTPCR negative for SARS-CoV-2 or could not be performed for any reason will be defined as probable COVID-19 case.

SECONDARY OUTCOMES:
Incidence of adverse drug reaction (ADR) | 4 weeks
  Any adverse reaction related to Hydroxychloroquine

CONTACTS AND LOCATIONS:
Overall Officials: Deba P Dhibar, MD, Principal Investigator — PGIMER, Chandigarh, India
Locations (2):
- India (2):
  - Post Graduate Institute of Medical Education and Research (PGIMER), Chandigarh
  - Post Graduate Institute of Medical Education and Research, Chandigarh

IPD SHARING:
Plan to Share IPD: No
Data will be shared with the concerned authority and Institutional Ethics committee as and when required.